CLINICAL TRIAL: NCT05941325
Title: Shanghai Sixth People's Hospital
Brief Title: A Single-arm, Open-label, Single-center Prospective Study of Fruquintinib Combined With Envafolimab in the Treatment of Advanced or Unresectable Locally Advanced Bone and Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Shuier Zheng, Director, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-025
Record Dates: First submitted 2023-06-28; First posted 2023-07-12 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Advanced or Unresectable Locally Advanced Bone and Soft Tissue Sarcoma
Keywords: fruquintinib; envafolimab; advanced or unresectable locally advanced bone and soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — HMPL-013; envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fruquintinib combined with envafolimab (Experimental)
  Interventions: Drug: fruquintinib; Drug: Envafolimab

INTERVENTIONS:
Drug: fruquintinib — VEGF receptor tyrosine-kinase inhibitor：fruquintinib（4mg), Oral，qd, d1-d14, Q3w，Until disease progression or intolerable toxicity occurs.
Drug: Envafolimab — anti-PD-1 immune checkpoint inhibitor：Envafolimab（400mg), subcutaneous injection, d1, Q3w，Until disease progression or intolerable toxicity occurs.

SUMMARY:
Many osteosarcomas are cured with a variety of combined chemotherapy and surgery, but a significant number will still relapse.VEGF promotes an immunosuppressive microenvironment and contributes to immune checkpoint inhibitor resistance in cancer.We aimed to explore the efficacy and safety of fruquintinib combined immunotherapy for bone and soft tissue sarcoma.

DETAILED DESCRIPTION:
A single-arm, open-label, single-center prospective study of fruquintinib combined with envafolimab in the treatment of advanced or unresectable locally advanced bone and soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* The subjects who volunteered to join the study signed the informed consent form, which showed good compliance and cooperated with the follow-up;
* 12-70 years old (boundary values included);
* Advanced or locally advanced bone and soft tissue sarcomas confirmed by histology or cytology, including but not limited to leiomyosarcomas, undifferentiated pleomorphic sarcomas, liposarcomas, synovial sarcomas, etc.;
* Patients with alveolar soft-tissue sarcoma, clear cell sarcoma, and other bone and soft-tissue sarcomas that progressed or recurred after at least previous anthracycline-containing chemotherapy regimens. Patients with bone and soft-tissue sarcoma who had not received previous first-line therapy were ineligible for chemotherapy or refused chemotherapy;
* At least one measurable lesion (RECIST 1.1);
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1 (amputation patients 0-2);
* Life expectancy > 12 weeks；
* Hematologic examination (no blood transfusion within 14 days):

  1. Neutrophil absolute value ≥1.5×109/L, platelet ≥100×109/L, hemoglobin concentration ≥9g/dL;
  2. Liver function (aspartate aminotransferase and glutamate aminotransferase ≤2.5×ULN, bilirubin ≤1.5×ULN; AST and ALT≤5×ULN if liver metastasis is present);
  3. Renal function (serum creatinine ≤1.5×ULN, or creatinine clearance rate (CCr)≥60ml/min);
  4. Coagulation, international standardized ratio (INR) ≤1.5, prothrombin time (PT) and activated partial thrombin time (APTT) ≤1.5×ULN;
  5. Thyroid function, thyroid stimulating hormone (TSH) ≤ the upper normal value (ULN); If abnormal, T3 and T4 levels should be examined, and if T3 and T4 levels are normal, they can be selected;
* Women of childbearing age must have taken a serum pregnancy test negative within 7 days prior to treatment and be willing to use medically approved effective contraception (e.g., an intrauterine device, contraceptive or condom) during the study period and for 3 months after the last study drug use; For male subjects whose partner is a woman of reproductive age, surgical sterilization is required or effective contraceptive methods are recommended during the study period and for 3 months after the last study treatment;
* The parents/guardians of the young patients have the ability to understand, agree to, and sign the study informed consent (ICF) prior to initiating any program-related procedures; Subject may give consent with parental/guardian consent (if applicable).

Exclusion Criteria:

* Had received radiotherapy for cancer, surgery, chemotherapy, immunotherapy, and other investigational drugs within 4 weeks prior to treatment;
* Previous treatment with anti-PD-1 or PD-L1 combined with anti-angiogenesis TKI;
* For soft tissue sarcomas, surgical and/or radiotherapy > 5% of the bone marrow area is planned during the study period;
* Had present central nervous system (CNS) metastases or prior brain metastases；
* Use of immunosuppressive drugs within 14 days prior to initiation of treatment, excluding transnasal and inhaled corticosteroids or physiological doses of systemic steroids (i.e., prednisolone dose not exceeding 10 mg per day or the physiological equivalent of other corticosteroids);
* History of any active autoimmune disease or autoimmune disease (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or asthma may have complete remission in childhood and do not currently require medical intervention or history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation);
* Severe infection (e.g., intravenous infusion of antibiotics, antifungals or antivirals) within 4 weeks prior to treatment, or unexplained fever >38.5 ℃ during screening/initial administration;
* Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal drug treatment);
* Significant clinical bleeding symptoms or significant bleeding tendency within 3 months prior to treatment (>30 ml within 3 months, appeared hematemesis, black dung, hematochezia) or hemoptysis (>5 mL of fresh blood within 4 weeks) , etc. Or treatment for venous/venous thrombosis events within the previous 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; Or long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day);
* Active heart disease, including myocardial infarction, severe/unstable angina within 6 months prior to treatment. Echocardiographic examination of left ventricular ejection fraction < 50%, poor arrhythmia control (including QTcF interval, men > 450 ms, female > 470 ms);
* Had other malignancies within the past 3 years or at the same time (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* Known to be allergic to the study drug or any of its excipients, or had severe allergic reactions to other monoclonal antibodies;
* Active or uncontrolled severe infection:

  1. Known human immunodeficiency virus (HIV) infection;
  2. A known history of clinically significant liver disease, including viral hepatitis [a known hepatitis B virus (HBV) carrier must exclude active HBV infection, i.e., positive HBV DNA (> 1×104 copies /mL or > 2000 IU/ mL);
  3. Known hepatitis C virus infection (HCV) with HCV RNA positive (> 1×103 copies /mL), or other hepatitis, cirrhosis];
* Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions which, according to judgement of the investigator, renders the patient inappropriate for using the investigational product or affect interpretation of study results;
* Urine routine indicates urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0 g.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | assessed up to 1 year
  The time from enrollment to disease progression or death.

SECONDARY OUTCOMES:
Overall Response Rate | assessed up to 1 year
  the proportion of patients with complete response and partial response , using RECIST v 1.1
Disease Control Rate | assessed up to 1 year
  the proportion of patients with complete response ，partial response and Stable Disease during or after treatment,using RECIST v 1.1
6-month Overall surviva | assessed up to 6 months
  time from date of enrolment to date of death of any reason within 6 months
overall survival rate | assessed up to 2 year
  time from date of enrolment to date of death of any reason.
Incidence of adverse events | assessed up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai No.6 People Hospital, Shanghai, Shanghai Municipality, China